CLINICAL TRIAL: NCT03509818
Title: Effects of the Physical Fitness on Serum Klotho Levels in Healthy Population: Response and Adaptation
Brief Title: Effects of the Physical Fitness on Serum Klotho Levels in Healthy Population
Acronym: CoFiKSa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Margarita Perez, Professor in Exercise Physiology, Universidad Europea de Madrid
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: Ref 47/764390.09/17
Record Dates: First submitted 2018-03-19; First posted 2018-04-26 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Healthy Population
Keywords: Klotho; Exercise; Physical Fitness
MeSH Terms: conditions — Motor Activity | interventions — Plyometric Exercise; Exercise

STUDY DESIGN:
Intervention Model Description: Description of the sample
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric (Experimental): Effects of plyometric acute exercise
  Interventions: Other: plyometric exercise
- Aerobic (Experimental): Effects of aerobic acute exercise
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: plyometric exercise — acute plyometric exercise
  Arms: Plyometric
Other: Aerobic exercise — acute aerobic exercise
  Arms: Aerobic

SUMMARY:
Exercise program in serum Klotho levels

DETAILED DESCRIPTION:
This study aims to analiyze the effects of acute exercise in serum Klotho levels attending physical fitness in healthy population

ELIGIBILITY:
Inclusion Criteria:

* healthy people between 20 and 45 years old

Exclusion Criteria:

* acute and chronic disease, people who take medication and supplements, smoker.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Change in serum Klotho levels | Baseline and one hour
  Change from baseline to acute exercise session

SECONDARY OUTCOMES:
Change in Cardiorespiratory Fitness VO2max | Baseline
  For this Variable All people Will perform a exercise test on treadmill (Tecnhogym run race 1400HC; Gambettola, Italy), in this way we determinate the VO2max. Through the modifies Balke protocol. The gas Exchange data Will measured breath by breath using open circuit spirometry and specific face mask for Fitmate, Cosmed; Vmax 29C, Sensormedics machine.
Change in Body Composition | Baseline
  The age in years; height in centimeters (tallimeter Ano Sayol SL, Barcelona, Spain); weight in kilograms (Inbody 720, Microcaya) and we can derive from this data the variable of Body Mass Index (BMI) calculated as weight (kg)/height (m2).
Change in Body Composition, Body muscle mass Index | Baseline
  For determinate this variable of the body composition will be use a Dual Densitometry X-Ray (DXA) (Hologic QDR Discovery, Bedford, MA, USA)
Change in Body Composition, % of Fat Mass | Baseline
  For determinate this variable of the body composition will be use a Dual Densitometry X-Ray (DXA) (Hologic QDR Discovery, Bedford, MA, USA)
Change in Body Composition, Total Muscle Mass | Baseline
  For determinate this variable of the body composition will be use a Dual Densitometry X-Ray (DXA) (Hologic QDR Discovery, Bedford, MA, USA)
Change in Body Composition, Visceral Fat Index. | Baseline
  For determinate this variable of the body composition will be use a Dual Densitometry X-Ray (DXA) (Hologic QDR Discovery, Bedford, MA, USA). This value is really important to determine a cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fernandez Elias, Ph, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Escuela de Doctorado e Invesitgacion, Universidad Europea, Madrid, Villaviciosa de Odon, Spain

IPD SHARING:
Plan to Share IPD: No